CLINICAL TRIAL: NCT00384930
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Design, 5-Group, Multinational Study to Evaluate the Efficacy, Dose Response, and Safety of Tadalafil Once-a-Day Dosing for 12 Weeks in Men With Signs and Symptoms of Benign Prostatic Hyperplasia
Brief Title: Study of Tadalafil Once-a Day for 12 Weeks in Men With Signs and Symptoms of Benign Prostatic Hyperplasia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: ICOS Corporation (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9797; H6D-MC-LVHG
Record Dates: First submitted 2006-10-03; First posted 2006-10-06 (Estimated); Results first posted 2009-08-19 (Estimated); Last update posted 2009-09-02 (Estimated); Status verified 2009-08

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Placebo Comparator): placebo tablet
  Interventions: Drug: placebo
- 2 (Active Comparator): 2.5 mg tadalafil tablet
  Interventions: Drug: tadalafil
- 3 (Active Comparator): 5 mg tadalafil tablet
  Interventions: Drug: tadalafil
- 4 (Active Comparator): 10 mg tadalafil tablet
  Interventions: Drug: tadalafil
- 5 (Active Comparator): 20 mg tadalafil tablet
  Interventions: Drug: tadalafil

INTERVENTIONS:
Drug: tadalafil — 2.5 mg tadalafil tablet by mouth once a day for twelve weeks.
  Other Names: LY450190; Cialis; IC351
  Arms: 2
Drug: tadalafil — 5 mg tadalafil tablet by mouth once a day for twelve weeks.
  Other Names: LY450190; Cialis; IC351
  Arms: 3
Drug: tadalafil — 10 mg tadalafil tablet by mouth once a day for twelve weeks.
  Other Names: LY450190; Cialis; IC351
  Arms: 4
Drug: tadalafil — 20 mg tadalafil tablet by mouth once a day for twelve weeks.
  Other Names: LY450190; Cialis; IC351
  Arms: 5
Drug: placebo — Placebo tablet taken by mouth one a day for twelve weeks
  Arms: 1

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel-design, multinational, 12-week study to compare the efficacy, dose response, and safety of tadalafil once a day versus placebo in men with signs and symptoms of benign prostatic hyperplasia, including lower urinary tract symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Males, 45 years or older, with benign prostatic hyperplasia, including lower urinary tract symptoms for at least 6 months prior to Visit 1 and an International Prostate Symptom Score (IPSS) greater than or equal to 13 at Visit 2.
* Agree not to use approved or experimental benign prostatic hyperplasia or erectile dysfunction treatments anytime during the study
* Have not taken finasteride or dutasteride therapy, any other lower urinary tract symptom (LUTS) therapy or phosphodiesterase type 5 (PDE5) inhibitors for specified duration of time prior to Visit 2.
* Have a prostate specific antigen (PSA) score within acceptable range defined for study or negative biopsy of the prostate for cancer within 12 months of Visit 1.

Exclusion Criteria:

* History of urinary retention or lower urinary tract (bladder) stones 6 months before the start of the study
* History of bladder outlet obstruction or urethral obstruction due to stricture, valves, sclerosis, or tumor.
* History of cardiac conditions including angina requiring certain treatment with nitrates, heart disease or coronary conditions including myocardial infarction, bypass surgery, angioplasty or stent placement for a specified time before starting the study.
* Certain neurological conditions associated with bladder problems or injuries to the brain or spinal cord within a specified time before starting the study.
* Nitrate use

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1058 (Actual)
Dates: Start 2006-08; Primary Completion 2007-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenwood, Indiana, United States

REFERENCES:
- [Derived] Vlachopoulos C, Oelke M, Maggi M, Mulhall JP, Rosenberg MT, Brock GB, Esler A, Buttner H. Impact of cardiovascular risk factors and related comorbid conditions and medical therapy reported at baseline on the treatment response to tadalafil 5 mg once-daily in men with lower urinary tract symptoms associated with benign prostatic hyperplasia: an integrated analysis of four randomised, double-blind, placebo-controlled, clinical trials. Int J Clin Pract. 2015 Dec;69(12):1496-507. doi: 10.1111/ijcp.12722. Epub 2015 Aug 24. PMID 26299520
- [Derived] Broderick GA, Brock GB, Roehrborn CG, Watts SD, Elion-Mboussa A, Viktrup L. Effects of tadalafil on lower urinary tract symptoms secondary to benign prostatic hyperplasia in men with or without erectile dysfunction. Urology. 2010 Jun;75(6):1452-8. doi: 10.1016/j.urology.2009.09.093. Epub 2010 Feb 16. PMID 20163842
- [Derived] Porst H, McVary KT, Montorsi F, Sutherland P, Elion-Mboussa A, Wolka AM, Viktrup L. Effects of once-daily tadalafil on erectile function in men with erectile dysfunction and signs and symptoms of benign prostatic hyperplasia. Eur Urol. 2009 Oct;56(4):727-35. doi: 10.1016/j.eururo.2009.04.033. Epub 2009 Apr 22. PMID 19409693
- [Derived] Roehrborn CG, McVary KT, Elion-Mboussa A, Viktrup L. Tadalafil administered once daily for lower urinary tract symptoms secondary to benign prostatic hyperplasia: a dose finding study. J Urol. 2008 Oct;180(4):1228-34. doi: 10.1016/j.juro.2008.06.079. Epub 2008 Aug 22. PMID 18722631
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Prior to randomization, participants had a 1-4 week Screening/Wash-out Period, followed by a 4 week Placebo Run-In Period. 1813 participants were screened with 755 screen failures, and 1058 participants randomized. The two participants who did not receive study drug were not included in the baseline demographics table.
Groups:
- Placebo: placebo tablet by mouth once a day for twelve weeks
- 2.5 mg Tadalafil: 2.5 mg tadalafil tablet by mouth once a day for twelve weeks
- 5 mg Tadalafil: 5 mg tadalafil tablet by mouth once a day for twelve weeks
- 10 mg Tadalafil: 10 mg tadalafil tablet by mouth once a day for twelve weeks
- 20 mg Tadalafil: 20 mg tadalafil tablet by mouth once a day for twelve weeks
Period: Overall Study
Arm/Group | Placebo | 2.5 mg Tadalafil | 5 mg Tadalafil | 10 mg Tadalafil | 20 mg Tadalafil
Started | 212 | 209 | 212 | 216 | 209
Received Double-Blind Study Drug | 211 | 208 | 212 | 216 | 209
Completed | 185 | 182 | 182 | 175 | 162
Not Completed | 27 | 27 | 30 | 41 | 47
Not completed — Adverse Event | 5 | 4 | 12 | 11 | 14
Not completed — Entry Criteria Not Met | 2 | 6 | 7 | 8 | 4
Not completed — Lack of Efficacy | 1 | 1 | 2 | 1 | 2
Not completed — Lost to Follow-up | 5 | 3 | 0 | 4 | 6
Not completed — Physician Decision | 0 | 1 | 1 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 1 | 6 | 4
Not completed — Sponsor Decision | 3 | 4 | 0 | 5 | 0
Not completed — Withdrawal by Subject | 9 | 7 | 7 | 6 | 16
Not completed — Didn't Receive Double-Blind Study Drug | 1 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 2.5 mg Tadalafil | 5 mg Tadalafil | 10 mg Tadalafil | 20 mg Tadalafil | Total
Number analyzed (Participants) | 211 | 208 | 212 | 216 | 209 | 1056
Age Continuous [Mean (Standard Deviation); unit: years] | 61.75 (7.69) | 62.03 (8.42) | 61.95 (8.17) | 62.22 (7.20) | 62.55 (8.09) | 62.10 (7.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 211 | 208 | 212 | 216 | 209 | 1056
Region of Enrollment [Number; unit: participants]
  Australia | 4 | 5 | 5 | 6 | 4 | 24
  Canada | 12 | 5 | 9 | 13 | 6 | 45
  France | 13 | 12 | 9 | 15 | 11 | 60
  Germany | 29 | 35 | 39 | 28 | 33 | 164
  Greece | 8 | 9 | 12 | 11 | 10 | 50
  Italy | 15 | 10 | 5 | 9 | 9 | 48
  Mexico | 19 | 16 | 17 | 19 | 19 | 90
  Spain | 3 | 3 | 2 | 5 | 4 | 17
  Sweden | 4 | 2 | 5 | 4 | 5 | 20
  United States | 105 | 112 | 109 | 106 | 108 | 540
Baseline (Visit 3) Lower Urinary Tract Symptoms (LUTS) Severity [Number; unit: participants] — LUTS Severity was measured with the International Prostate Symptom Score (IPSS), which has a scoring range of 0 to 35. Total scores: 0-7 Mildly symptomatic; 8-19 moderately symptomatic; 20-35 severely symptomatic.
  participants
    Moderate (<20 units on a scale: IPSS) | 137 | 139 | 141 | 143 | 141 | 701
    Severe (>=20 units on a scale: IPSS) | 74 | 69 | 71 | 72 | 68 | 354
    Unknown | 0 | 0 | 0 | 1 | 0 | 1
Duration of Lower Urinary Tract Symptoms (LUTS) Secondary to Benign Prostatic Hyperplasia (BPH) [Number; unit: participants]
  < 6 months | 0 | 0 | 0 | 1 | 0 | 1
  6 months to 1 year | 44 | 27 | 37 | 27 | 39 | 174
  1 year to 3 years | 62 | 64 | 63 | 81 | 70 | 340
  > 3 years | 105 | 117 | 112 | 107 | 100 | 541
Erectile Dysfunction [Number; unit: participants]
  Yes | 142 | 135 | 144 | 150 | 145 | 716
  No | 67 | 71 | 68 | 64 | 61 | 331
  Unknown | 1 | 2 | 0 | 2 | 3 | 8
  Not Collected | 1 | 0 | 0 | 0 | 0 | 1
Previous Therapy for Benign Prostatic Hyperplasia (BPH) [Number; unit: participants]
  No | 153 | 139 | 158 | 160 | 152 | 762
  Yes | 58 | 69 | 54 | 56 | 57 | 294
Race/Ethnicity [Number; unit: participants]
  African | 3 | 3 | 7 | 5 | 5 | 23
  Caucasian | 179 | 184 | 179 | 186 | 176 | 904
  East Asian | 0 | 1 | 1 | 0 | 0 | 2
  Hispanic | 29 | 20 | 25 | 24 | 25 | 123
  West Asian | 0 | 0 | 0 | 1 | 3 | 4
Severity of Erectile Dysfunction (ED) [Number; unit: participants] — Severity was determine only on participants with Erectile Dysfunction using scores on International Index of Erectile Function (IIEF) EF Domain (sum of the scores for Questions 1 through 5 and Question 15) with a range of 0 to 30. Normal EF (≥26), mild ED (17 to 25), moderate ED (11 to 16), and severe ED (1 to 10).
  participants
    Mild | 38 | 42 | 41 | 56 | 40 | 217
    Moderate | 82 | 75 | 82 | 72 | 79 | 390
    Severe | 22 | 18 | 21 | 22 | 26 | 109
Sexually Active [Number; unit: participants]
  No | 42 | 40 | 33 | 42 | 48 | 205
  Yes | 169 | 168 | 179 | 174 | 161 | 851
Sexually Active and Erectile Dysfunction (ED) [Number; unit: participants]
  Sexually Active with ED | 115 | 113 | 117 | 120 | 116 | 581
  Sexually Active without ED | 54 | 55 | 62 | 54 | 45 | 270
  Not Sexually Active with ED | 26 | 21 | 25 | 28 | 28 | 128
  Not Sexually Active without ED | 15 | 17 | 8 | 12 | 18 | 70
  Sexual Activity and/or ED Status is Unknown | 1 | 2 | 0 | 2 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 12 Week Endpoint in International Prostate Symptom Score (IPSS): Primary Analysis
Description: Assesses the severity of BPH-LUTS and the response to therapy. The total score was derived by summing the scores of the responses to the 7 component questions. Scores range from 0 to 35; 0-7 Mildly symptomatic; 8-19 moderately symptomatic; 20-35 severely symptomatic.
Time Frame: Baseline and 12 weeks
Population: Primary analysis was performed on an intent-to-treat basis. Data from subjects with baseline and at least one postbaseline were used for the analysis. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: placebo tablet taken by mouth once a day for 12 weeks
- 5 mg Tadalafil: 5 mg tadalafil tablet taken by mouth once a day for 12 weeks
Arm/Group | Placebo | 5 mg Tadalafil
Number analyzed (Participants) | 205 | 205
units on a scale
  Baseline | 17.08 (6.36) | 17.30 (5.97)
  Change from Baseline | -2.25 (6.17) | -4.92 (5.67)
Statistical Analysis 1: Comparison: Placebo vs 5 mg Tadalafil; This is the principal inferential analysis of the primary outcome; Test type: Superiority or Other; p < 0.001, Permutation Test — P-value for Change from Baseline. Change = Endpoint minus Baseline

2. Secondary Outcome: Change From Baseline to 12 Week Endpoint in International Prostate Symptom Score (IPSS) (Irritative) Subscore
Description: Measures irritative symptoms over the past 4 weeks of the IPSS. IPSS irritative subscore is the sum of Questions 2, 4 and 7 of the IPSS questionnaire. Scores range from 1 (few irritative symptoms) to 5 (frequent irritative symptoms), thus the 3 questions of the irritative subscore range from 0 to 15.
Time Frame: baseline and 12 weeks
Population: Secondary continuous analyses were performed on an intent-to-treat basis. Data from subjects with baseline and at least one postbaseline were used for the analysis. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 2.5 mg Tadalafil | 5 mg Tadalafil | 10 mg Tadalafil | 20 mg Tadalafil
Number analyzed (Participants) | 205 | 201 | 205 | 208 | 199
units on a scale
  Baseline | 7.58 (3.09) | 7.78 (2.86) | 7.65 (2.84) | 7.88 (2.67) | 7.53 (3.07)
  Change from Baseline | -0.99 (2.92) | -1.62 (2.83) | -1.91 (2.64) | -2.04 (2.75) | -2.05 (2.86)
Statistical Analysis 1: Comparison: Placebo vs 2.5 mg Tadalafil; Test type: Superiority or Other; p = 0.025, ANCOVA — P-value for Change from Baseline. Change=Endpoint - Baseline. P-values from ANCOVA model with effect of treatment group, geographic region, and baseline value of analyzed variable as a covariate, and were not adjusted for multiple comparisons; Mean Difference (Net) = -0.57, 95% CI [-1.08 to -0.07] — Mean Difference = 2.5 mg Tadalafil minus Placebo
Statistical Analysis 2: Comparison: Placebo vs 5 mg Tadalafil; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.90, 95% CI [-1.40 to -0.40] — Mean Difference = 5 mg Tadalafil minus Placebo
Statistical Analysis 3: Comparison: Placebo vs 10 mg Tadalafil; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.96, 95% CI [-1.45 to -0.46] — Mean Difference = 10 mg Tadalafil minus Placebo
Statistical Analysis 4: Comparison: Placebo vs 20 mg Tadalafil; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -1.07, 95% CI [-1.58 to -0.57] — Mean Difference = 20 mg Tadalafil minus Placebo

3. Secondary Outcome: Change From Baseline to 12 Week Endpoint in International Prostate Symptom Score (IPSS) Voiding (Obstructive) Subscore
Description: Measures obstructive symptoms over the past 4 weeks of the IPSS. IPSS obstructive subscore is the sum of Questions 1, 3, 5 and 6 of the IPSS questionnaire. Scores range from 1 (few obstructive symptoms) to 5 (frequent obstructive symptoms), thus the 4 questions of the obstructive score range from 0 to 20.
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 2.5 mg Tadalafil | 5 mg Tadalafil | 10 mg Tadalafil | 20 mg Tadalafil
Number analyzed (Participants) | 205 | 202 | 205 | 207 | 199
units on a scale
  Baseline | 9.51 (4.21) | 9.71 (4.16) | 9.65 (4.10) | 9.88 (3.87) | 9.57 (4.45)
  Change from Baseline | -1.27 (4.00) | -2.31 (3.84) | -3.00 (3.87) | -3.29 (4.04) | -3.17 (4.02)
Statistical Analysis 1: Comparison: Placebo vs 2.5 mg Tadalafil; Test type: Superiority or Other; p = 0.008, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.97, 95% CI [-1.69 to -0.26] — Mean Difference = 2.5 mg Tadalafil minus Placebo
Statistical Analysis 2: Comparison: Placebo vs 5 mg Tadalafil; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -1.69, 95% CI [-2.40 to -0.98] — Mean Difference = 5 mg Tadalafil minus Placebo
Statistical Analysis 3: Comparison: Placebo vs 10 mg Tadalafil; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -1.89, 95% CI [-2.60 to -1.18] — Mean Difference = 10 mg Tadalafil minus Placebo
Statistical Analysis 4: Comparison: Placebo vs 20 mg Tadalafil; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -1.87, 95% CI [-2.59 to -1.15] — Mean Difference = 20 mg Tadalafil minus Placebo

4. Secondary Outcome: Change From Baseline to 12 Week Endpoint in International Prostate Symptom Score (IPSS) Question 7 (Nocturia)
Description: Measures nocturia (the need to get up at night to urinate) over the past 4 weeks. Scores range from 1 (few episodes of nocturia) to 5 (frequent episodes of nocturia).
Time Frame: baseline and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 2.5 mg Tadalafil | 5 mg Tadalafil | 10 mg Tadalafil | 20 mg Tadalafil
Number analyzed (Participants) | 205 | 201 | 205 | 208 | 199
units on a scale
  Baseline | 2.36 (1.10) | 2.37 (1.31) | 2.36 (1.91) | 2.36 (1.15) | 2.20 (1.23)
  Change from Baseline | -0.36 (1.09) | -0.43 (1.33) | -0.49 (1.17) | -0.43 (1.28) | -0.54 (1.17)
Statistical Analysis 1: Comparison: Placebo vs 2.5 mg Tadalafil; Test type: Superiority or Other; p = 0.503, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.07, 95% CI [-0.28 to 0.14] — Mean Difference = 2.5 mg Tadalafil minus Placebo
Statistical Analysis 2: Comparison: Placebo vs 5 mg Tadalafil; Test type: Superiority or Other; p = 0.206, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.13, 95% CI [-0.34 to 0.07] — Mean Difference = 5 mg Tadalafil minus Placebo
Statistical Analysis 3: Comparison: Placebo vs 10 mg Tadalafil; Test type: Superiority or Other; p = 0.452, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.08, 95% CI [-0.28 to 0.13] — Mean Difference = 10 mg Tadalafil minus Placebo
Statistical Analysis 4: Comparison: Placebo vs 20 mg Tadalafil; Test type: Superiority or Other; p = 0.012, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.26, 95% CI [-0.47 to -0.06] — Mean Difference = 20 mg Tadalafil minus Placebo

5. Secondary Outcome: Change From Baseline to 12 Week Endpoint in International Prostate Symptom Score (IPSS) Quality of Life (QoL) Index
Description: Assessment of quality of life (QOL) by urinary symptoms, with scores ranging from 0 (delighted) to 6 (terrible).
Time Frame: baseline and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 5.0 mg Tadalafil: 5.0 mg tadalafil tablet by mouth once a day for twelve weeks
Arm/Group | Placebo | 2.5 mg Tadalafil | 5.0 mg Tadalafil | 10 mg Tadalafil | 20 mg Tadalafil
Number analyzed (Participants) | 205 | 202 | 205 | 206 | 199
units on a scale
  Baseline | 3.57 (1.19) | 3.69 (1.19) | 3.54 (1.30) | 3.55 (1.23) | 3.59 (1.28)
  Change from Baseline | -0.56 (1.20) | -0.86 (1.13) | -0.92 (1.30) | -0.98 (1.46) | -0.97 (1.27)
Statistical Analysis 1: Comparison: Placebo vs 2.5 mg Tadalafil; Test type: Superiority or Other; p = 0.029, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.26, 95% CI [-0.49 to -0.03] — Mean Difference = 2.5 mg Tadalafil minus Placebo
Statistical Analysis 2: Comparison: Placebo vs 5.0 mg Tadalafil; Test type: Superiority or Other; p = 0.002, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.37, 95% CI [-0.60 to -0.14] — Mean Difference = 5 mg Tadalafil minus Placebo
Statistical Analysis 3: Comparison: Placebo vs 10 mg Tadalafil; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.43, 95% CI [-0.66 to -0.19] — Mean Difference = 10 mg Tadalafil minus Placebo
Statistical Analysis 4: Comparison: Placebo vs 20 mg Tadalafil; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.40, 95% CI [-0.64 to -0.17] — Mean Difference = 20 mg Tadalafil minus Placebo

6. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Benign Prostatic Hyperplasia Impact Index (BII)
Description: Measures the impact that symptoms of BPH has on the patients well being. This questionnaire has 4 questions assessing the level of urinary discomfort and it's impact on the patients. Three questions range from 0 (no impact) to 4 (high impact); one question ranges from 0 (low impact) to 4 (high impact). The BII score ranges from 0 to 16.
Time Frame: baseline and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 2.5 mg Tadalafil | 5 mg Tadalafil | 10 mg Tadalafil | 20 mg Tadalafil
Number analyzed (Participants) | 205 | 201 | 204 | 209 | 199
units on a scale
  Baseline | 4.94 (2.95) | 4.73 (2.95) | 4.66 (2.98) | 4.86 (2.98) | 4.75 (2.79)
  Change from Baseline | -0.79 (2.52) | -0.83 (2.66) | -1.25 (2.75) | -1.31 (2.79) | -1.34 (2.41)
Statistical Analysis 1: Comparison: Placebo vs 2.5 mg Tadalafil; Test type: Superiority or Other; p = 0.583, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.13, 95% CI [-0.58 to 0.33] — Mean Difference = 2.5 mg Tadalafil minus Placebo
Statistical Analysis 2: Comparison: Placebo vs 5 mg Tadalafil; Test type: Superiority or Other; p = 0.013, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.57, 95% CI [-1.03 to -0.12] — Mean Difference = 5 mg Tadalafil minus Placebo
Statistical Analysis 3: Comparison: Placebo vs 10 mg Tadalafil; Test type: Superiority or Other; p = 0.016, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.55, 95% CI [-1.00 to -0.10] — Mean Difference = 10 mg Tadalafil minus Placebo
Statistical Analysis 4: Comparison: Placebo vs 20 mg Tadalafil; Test type: Superiority or Other; p = 0.007, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.62, 95% CI [-1.08 to -0.17] — Mean Difference = 20 mg Tadalafil minus Placebo

7. Secondary Outcome: Number of Participants Who Answer "Yes" to the Lower Urinary Tract Symptoms (LUTS) Global Assessment Question (LUTS-GAQ)
Description: LUTS-GAQ Question asks the participant if the treatment they have been on has improved their uninary symptoms.
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Placebo | 2.5 mg Tadalafil | 5 mg Tadalafil | 10 mg Tadalafil | 20 mg Tadalafil
Number analyzed (Participants) | 199 | 194 | 201 | 200 | 186
participants | 109 | 120 | 139 | 146 | 138
Statistical Analysis 1: Comparison: Placebo vs 2.5 mg Tadalafil; Test type: Superiority or Other; p = 0.133, Cochran-Mantel-Haenszel — P-values are from Cochran-Mantel-Haenszel test stratified by the randomization strata factors (4 geographic regions, 2 levels of IPSS severity, 2 levels of ED history) as fixed effect, and were not adjusted for multiple comparisons
Statistical Analysis 2: Comparison: Placebo vs 5 mg Tadalafil; Test type: Superiority or Other; p = 0.003, Cochran-Mantel-Haenszel — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs 10 mg Tadalafil; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs 20 mg Tadalafil; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 7, analysis 1]

8. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Peak Urinary Flow
Description: Measures the maximum flow rate of urine (measured in mL/s). This is a continuous parameter with positive numeric values.
Time Frame: baseline and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milliliter per second
Arm/Group | Placebo | 2.5 mg Tadalafil | 5 mg Tadalafil | 10 mg Tadalafil | 20 mg Tadalafil
Number analyzed (Participants) | 198 | 201 | 202 | 201 | 190
milliliter per second
  Baseline | 10.31 (4.85) | 9.97 (4.09) | 10.37 (3.86) | 9.93 (3.77) | 9.82 (3.97)
  Change from Baseline | 1.23 (5.01) | 1.50 (4.56) | 1.61 (3.95) | 1.69 (4.46) | 2.15 (4.69)
Statistical Analysis 1: Comparison: Placebo vs 2.5 mg Tadalafil; Test type: Superiority or Other; p = 0.735, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.14, 95% CI [-0.69 to 0.98] — Mean Difference = 2.5 mg Tadalafil minus Placebo
Statistical Analysis 2: Comparison: Placebo vs 5 mg Tadalafil; Test type: Superiority or Other; p = 0.355, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.39, 95% CI [-0.44 to 1.23] — Mean Difference = 5 mg Tadalafil minus Placebo
Statistical Analysis 3: Comparison: Placebo vs 10 mg Tadalafil; Test type: Superiority or Other; p = 0.433, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.34, 95% CI [-0.50 to 1.17] — Mean Difference = 10 mg Tadalafil minus Placebo
Statistical Analysis 4: Comparison: Placebo vs 20 mg Tadalafil; Test type: Superiority or Other; p = 0.089, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.74, 95% CI [-0.11 to 1.59] — Mean Difference = 20 mg Tadalafil minus Placebo

9. Secondary Outcome: Change From Baseline to 12 Week Endpoint in International Index of Erectile Function (IIEF) EF Domain
Description: Measures erectile function over the past 4 weeks on Questions 1-5 and 15 (6 questions) of the International Index of Erecile Function (IIEF) questionnaire. Scores range from 0 (low/no erectile function) to 5 (high erectile function), thus the 6 questions of the IIEF-EF domain range from 0 to 30.
Time Frame: baseline and 12 weeks
Population: Secondary continuous analyses were performed on an intent-to-treat basis. Data from all randomized and sexually active subjects with a history of ED and non-missing data at baseline and at least one postbaseline visit were used for the analysis. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 2.5 mg Tadalafil | 5 mg Tadalafil | 10 mg Tadalafil | 20 mg Tadalafil
Number analyzed (Participants) | 113 | 109 | 113 | 113 | 109
units on a scale
  Baseline | 17.26 (7.95) | 17.42 (8.30) | 15.29 (8.13) | 17.22 (8.43) | 16.28 (8.05)
  Change from Baseline | 0.78 (6.32) | 3.97 (7.30) | 6.56 (9.43) | 6.64 (8.29) | 7.44 (8.42)
Statistical Analysis 1: Comparison: Placebo vs 2.5 mg Tadalafil; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 3.36, 95% CI [1.56 to 5.17] — Mean Difference = 2.5 mg Tadalafil minus Placebo
Statistical Analysis 2: Comparison: Placebo vs 5 mg Tadalafil; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 4.75, 95% CI [2.95 to 6.54] — Mean Difference = 5 mg Tadalafil minus Placebo
Statistical Analysis 3: Comparison: Placebo vs 10 mg Tadalafil; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 5.83, 95% CI [4.04 to 7.62] — Mean Difference = 10 mg Tadalafil minus Placebo
Statistical Analysis 4: Comparison: Placebo vs 20 mg Tadalafil; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 6.15, 95% CI [4.35 to 7.95] — Mean Difference = 20 mg Tadalafil minus Placebo

10. Primary Outcome: Change From Baseline to Week 12 in International Prostate Symptom Score (IPSS): Supportive Analysis
Description: as for outcome 1
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 2.5 mg Tadalafil | 5 mg Tadalafil | 10 mg Tadalafil | 20 mg Tadalafil
Number analyzed (Participants) | 205 | 201 | 205 | 207 | 199
units on a scale | -2.23 (0.49) | -3.81 (0.50) | -4.83 (0.49) | -5.13 (0.48) | -5.17 (0.50)
Statistical Analysis 1: Comparison: Placebo vs 2.5 mg Tadalafil; This is a supportive analysis of the primary outcome; Test type: Superiority or Other; p = 0.005, ANCOVA — P-values are from an ANCOVA model with effect of treatment group, geographic region, and IPSS baseline value (at Visit 3) as a covariate, and were not adjusted for multiple comparisons; Mean Difference (Net) = -1.58, 95% CI [-2.68 to -0.48] — Mean Difference = 2.5 mg Tadalafil minus Placebo
Statistical Analysis 2: Comparison: Placebo vs 5 mg Tadalafil; This is a supportive analysis of the primary outcome; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Mean Difference (Net) = -2.60, 95% CI [-3.69 to -1.51] — Mean Difference = 5 mg Tadalafil minus Placebo
Statistical Analysis 3: Comparison: Placebo vs 10 mg Tadalafil; This is a supportive analysis of the primary outcome; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Mean Difference (Net) = -2.90, 95% CI [-3.99 to -1.81] — Mean Difference = 10 mg Tadalafil minus Placebo
Statistical Analysis 4: Comparison: Placebo vs 20 mg Tadalafil; This is a supportive analysis of the primary outcome; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Mean Difference (Net) = -2.94, 95% CI [-4.04 to -1.84] — Mean Difference = 20 mg Tadalafil minus Placebo

ADVERSE EVENTS:
Arm/Group | Placebo | 2.5 mg Tadalafil | 5 mg Tadalafil | 10 mg Tadalafil | 20 mg Tadalafil
Serious Adverse Events (participants affected / at risk) | 6 | 3 | 1 | 2 | 5
Other Adverse Events (participants affected / at risk) | 43 | 54 | 65 | 75 | 80
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Placebo | 2.5 mg Tadalafil | 5 mg Tadalafil | 10 mg Tadalafil | 20 mg Tadalafil
Angina unstable (Cardiac disorders) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 1/216 (1) | 0/209 (0)
Atrial tachycardia (Cardiac disorders) | 0/212 (0) | 1/209 (1) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Coronary artery stenosis (Cardiac disorders) | 1/212 (1) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Myocardial infarction (Cardiac disorders) | 0/212 (0) | 1/209 (1) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Pancreatitis (Gastrointestinal disorders) | 0/212 (0) | 0/209 (0) | 1/212 (1) | 0/216 (0) | 0/209 (0)
Cholecystitis (Hepatobiliary disorders) | 0/212 (0) | 0/209 (0) | 1/212 (1) | 0/216 (0) | 0/209 (0)
Cartilage injury (Injury, poisoning and procedural complications) | 1/212 (1) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1/212 (1) | 0/209 (0) | 0/212 (0) | 1/216 (1) | 1/209 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 1/209 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1/212 (1) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1/212 (2) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/212 (0) | 1/209 (1) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Cerebrovascular accident (Nervous system disorders) | 1/212 (1) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 1/209 (1)
Nephrolithiasis (Renal and urinary disorders) | 0/212 (0) | 1/209 (1) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Renal colic (Renal and urinary disorders) | 1/212 (1) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Renal failure acute (Renal and urinary disorders) | 0/212 (0) | 1/209 (1) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Ureteric rupture (Renal and urinary disorders) | 0/212 (0) | 1/209 (1) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Urinary retention (Renal and urinary disorders) | 1/212 (1) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 1/209 (1)
Coronary arterial stent insertion (Surgical and medical procedures) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 1/209 (1)
Indwelling catheter management (Surgical and medical procedures) | 1/212 (1) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Ureteral catheterisation (Surgical and medical procedures) | 1/212 (1) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Ureteral stent insertion (Surgical and medical procedures) | 0/212 (0) | 1/209 (1) | 0/212 (0) | 0/216 (0) | 0/209 (0)
OTHER ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Placebo | 2.5 mg Tadalafil | 5 mg Tadalafil | 10 mg Tadalafil | 20 mg Tadalafil
Arrhythmia (Cardiac disorders) | 0/212 (0) | 1/209 (1) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Atrioventricular block second degree (Cardiac disorders) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 1/209 (1)
Cardiomegaly (Cardiac disorders) | 0/212 (0) | 0/209 (0) | 1/212 (1) | 0/216 (0) | 0/209 (0)
Left atrial dilatation (Cardiac disorders) | 1/212 (1) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Sinus arrhythmia (Cardiac disorders) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 1/209 (1)
Tachycardia (Cardiac disorders) | 0/212 (0) | 0/209 (0) | 1/212 (1) | 0/216 (0) | 1/209 (1)
Ear congestion (Ear and labyrinth disorders) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 1/216 (1) | 0/209 (0)
Ear pain (Ear and labyrinth disorders) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 1/209 (1)
Tinnitus (Ear and labyrinth disorders) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 1/216 (1) | 0/209 (0)
Vertigo (Ear and labyrinth disorders) | 0/212 (0) | 0/209 (0) | 1/212 (2) | 0/216 (0) | 1/209 (1)
Hypothyroidism (Endocrine disorders) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 1/209 (1)
Choroidal neovascularisation (Eye disorders) | 0/212 (0) | 0/209 (0) | 1/212 (1) | 0/216 (0) | 0/209 (0)
Conjunctivitis (Eye disorders) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 1/209 (1)
Eye irritation (Eye disorders) | 0/212 (0) | 0/209 (0) | 1/212 (1) | 0/216 (0) | 1/209 (1)
Eye pain (Eye disorders) | 1/212 (1) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Eyelid irritation (Eye disorders) | 1/212 (1) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Glaucoma (Eye disorders) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 1/216 (1) | 0/209 (0)
Ocular hyperaemia (Eye disorders) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 1/209 (1)
Ocular hypertension (Eye disorders) | 0/212 (0) | 0/209 (0) | 1/212 (1) | 0/216 (0) | 0/209 (0)
Panophthalmitis (Eye disorders) | 1/212 (2) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Photopsia (Eye disorders) | 0/212 (0) | 0/209 (0) | 1/212 (1) | 0/216 (0) | 0/209 (0)
Retinal tear (Eye disorders) | 0/212 (0) | 0/209 (0) | 1/212 (2) | 0/216 (0) | 0/209 (0)
Vision blurred (Eye disorders) | 1/212 (1) | 0/209 (0) | 1/212 (1) | 0/216 (0) | 0/209 (0)
Vitreous floaters (Eye disorders) | 0/212 (0) | 0/209 (0) | 1/212 (1) | 0/216 (0) | 0/209 (0)
Abdominal pain (Gastrointestinal disorders) | 0/212 (0) | 1/209 (1) | 1/212 (1) | 1/216 (1) | 1/209 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0/212 (0) | 1/209 (1) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2/212 (2) | 2/209 (3) | 2/212 (2) | 3/216 (3) | 0/209 (0)
Bowel movement irregularity (Gastrointestinal disorders) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 1/209 (1)
Constipation (Gastrointestinal disorders) | 1/212 (1) | 0/209 (0) | 0/212 (0) | 1/216 (1) | 0/209 (0)
Diarrhoea (Gastrointestinal disorders) | 3/212 (3) | 2/209 (2) | 6/212 (12) | 1/216 (1) | 5/209 (5)
Duodenogastric reflux (Gastrointestinal disorders) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 1/209 (1)
Dyspepsia (Gastrointestinal disorders) | 0/212 (0) | 2/209 (3) | 10/212 (15) | 6/216 (6) | 10/209 (10)
Flatulence (Gastrointestinal disorders) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 1/216 (1) | 1/209 (1)
Gastritis (Gastrointestinal disorders) | 1/212 (1) | 0/209 (0) | 1/212 (1) | 3/216 (3) | 2/209 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0/212 (0) | 2/209 (2) | 2/212 (2) | 6/216 (6) | 3/209 (3)
Gingival disorder (Gastrointestinal disorders) | 0/212 (0) | 1/209 (1) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Haemorrhoids (Gastrointestinal disorders) | 1/212 (1) | 1/209 (1) | 0/212 (0) | 1/216 (1) | 0/209 (0)
Hiatus hernia (Gastrointestinal disorders) | 0/212 (0) | 1/209 (1) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Inguinal hernia (Gastrointestinal disorders) | 0/212 (0) | 0/209 (0) | 1/212 (1) | 0/216 (0) | 0/209 (0)
Nausea (Gastrointestinal disorders) | 1/212 (1) | 0/209 (0) | 3/212 (3) | 0/216 (0) | 0/209 (0)
Oesophageal pain (Gastrointestinal disorders) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 1/216 (1) | 0/209 (0)
Oesophagitis (Gastrointestinal disorders) | 0/212 (0) | 1/209 (1) | 0/212 (0) | 0/216 (0) | 1/209 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0/212 (0) | 0/209 (0) | 1/212 (1) | 0/216 (0) | 0/209 (0)
Reflux oesophagitis (Gastrointestinal disorders) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 1/216 (1) | 1/209 (1)
Stomach discomfort (Gastrointestinal disorders) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 1/209 (1)
Tooth loss (Gastrointestinal disorders) | 0/212 (0) | 0/209 (0) | 1/212 (1) | 0/216 (0) | 0/209 (0)
Toothache (Gastrointestinal disorders) | 0/212 (0) | 1/209 (1) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Vomiting (Gastrointestinal disorders) | 1/212 (1) | 0/209 (0) | 3/212 (3) | 0/216 (0) | 1/209 (1)
Asthenia (General disorders) | 1/212 (1) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 1/209 (1)
Chest discomfort (General disorders) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 1/209 (1)
Chest pain (General disorders) | 0/212 (0) | 0/209 (0) | 3/212 (3) | 0/216 (0) | 0/209 (0)
Fatigue (General disorders) | 1/212 (1) | 0/209 (0) | 1/212 (1) | 1/216 (1) | 0/209 (0)
Inflammation (General disorders) | 0/212 (0) | 0/209 (0) | 1/212 (1) | 0/216 (0) | 0/209 (0)
Influenza like illness (General disorders) | 0/212 (0) | 0/209 (0) | 1/212 (1) | 0/216 (0) | 0/209 (0)
Irritability (General disorders) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 1/216 (1) | 0/209 (0)
Local swelling (General disorders) | 0/212 (0) | 1/209 (1) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Oedema (General disorders) | 0/212 (0) | 0/209 (0) | 1/212 (1) | 1/216 (1) | 0/209 (0)
Oedema peripheral (General disorders) | 0/212 (0) | 1/209 (1) | 1/212 (1) | 2/216 (2) | 0/209 (0)
Pain (General disorders) | 0/212 (0) | 1/209 (1) | 2/212 (2) | 0/216 (0) | 1/209 (1)
Pyrexia (General disorders) | 1/212 (1) | 0/209 (0) | 2/212 (2) | 0/216 (0) | 1/209 (1)
Sensation of foreign body (General disorders) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 2/209 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 1/212 (1) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Hypersensitivity (Immune system disorders) | 0/212 (0) | 0/209 (0) | 1/212 (1) | 0/216 (0) | 1/209 (1)
Seasonal allergy (Immune system disorders) | 0/212 (0) | 0/209 (0) | 1/212 (2) | 0/216 (0) | 1/209 (1)
Bronchitis (Infections and infestations) | 1/212 (1) | 3/209 (3) | 1/212 (1) | 5/216 (5) | 0/209 (0)
Cystitis (Infections and infestations) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 1/209 (1)
Diverticulitis (Infections and infestations) | 0/212 (0) | 1/209 (1) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Ear infection (Infections and infestations) | 0/212 (0) | 0/209 (0) | 1/212 (1) | 0/216 (0) | 0/209 (0)
Folliculitis (Infections and infestations) | 0/212 (0) | 1/209 (1) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Fungal infection (Infections and infestations) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 1/216 (1) | 0/209 (0)
Gastroenteritis (Infections and infestations) | 0/212 (0) | 1/209 (1) | 0/212 (0) | 1/216 (1) | 0/209 (0)
Gastroenteritis viral (Infections and infestations) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 2/216 (2) | 1/209 (1)
Herpes simplex (Infections and infestations) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 1/209 (1)
Herpes zoster (Infections and infestations) | 1/212 (1) | 1/209 (1) | 0/212 (0) | 0/216 (0) | 2/209 (2)
Influenza (Infections and infestations) | 1/212 (1) | 4/209 (4) | 4/212 (4) | 1/216 (1) | 2/209 (2)
Labyrinthitis (Infections and infestations) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 1/216 (1) | 0/209 (0)
Lower respiratory tract infection (Infections and infestations) | 1/212 (1) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Nasopharyngitis (Infections and infestations) | 2/212 (2) | 7/209 (8) | 4/212 (6) | 2/216 (2) | 5/209 (5)
Pharyngitis (Infections and infestations) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 2/216 (2) | 0/209 (0)
Pneumonia viral (Infections and infestations) | 0/212 (0) | 0/209 (0) | 1/212 (1) | 0/216 (0) | 0/209 (0)
Rhinitis (Infections and infestations) | 0/212 (0) | 0/209 (0) | 1/212 (1) | 0/216 (0) | 0/209 (0)
Sinusitis (Infections and infestations) | 1/212 (1) | 1/209 (1) | 0/212 (0) | 1/216 (1) | 1/209 (1)
Tooth abscess (Infections and infestations) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 1/216 (1) | 0/209 (0)
Tracheitis (Infections and infestations) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 1/216 (1) | 0/209 (0)
Upper respiratory tract infection (Infections and infestations) | 2/212 (2) | 0/209 (0) | 2/212 (2) | 0/216 (0) | 1/209 (1)
Urinary tract infection (Infections and infestations) | 3/212 (3) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Animal bite (Injury, poisoning and procedural complications) | 1/212 (1) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Back injury (Injury, poisoning and procedural complications) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 1/216 (1) | 1/209 (1)
Excoriation (Injury, poisoning and procedural complications) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 1/216 (1) | 0/209 (0)
Fall (Injury, poisoning and procedural complications) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 1/216 (1) | 0/209 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1/212 (1) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Joint sprain (Injury, poisoning and procedural complications) | 0/212 (0) | 2/209 (2) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 1/209 (1)
Limb injury (Injury, poisoning and procedural complications) | 1/212 (1) | 0/209 (0) | 0/212 (0) | 1/216 (1) | 0/209 (0)
Skeletal injury (Injury, poisoning and procedural complications) | 0/212 (0) | 0/209 (0) | 1/212 (1) | 0/216 (0) | 0/209 (0)
Tendon injury (Injury, poisoning and procedural complications) | 0/212 (0) | 0/209 (0) | 1/212 (1) | 0/216 (0) | 0/209 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 1/216 (1) | 0/209 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0/212 (0) | 1/209 (1) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Vertebral injury (Injury, poisoning and procedural complications) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 1/216 (1) | 0/209 (0)
Wound (Injury, poisoning and procedural complications) | 0/212 (0) | 0/209 (0) | 1/212 (2) | 0/216 (0) | 0/209 (0)
Arthroscopy (Investigations) | 1/212 (1) | 0/209 (0) | 0/212 (0) | 1/216 (1) | 0/209 (0)
Blood creatine phosphokinase increased (Investigations) | 0/212 (0) | 1/209 (1) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Cardiac murmur (Investigations) | 1/212 (1) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Gamma-glutamyltransferase increased (Investigations) | 1/212 (1) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Heart rate abnormal (Investigations) | 0/212 (0) | 1/209 (1) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Heart rate irregular (Investigations) | 0/212 (0) | 1/209 (2) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Hepatic enzyme increased (Investigations) | 1/212 (1) | 0/209 (0) | 1/212 (1) | 0/216 (0) | 0/209 (0)
Prostatic specific antigen increased (Investigations) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 1/216 (1) | 0/209 (0)
Weight increased (Investigations) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 1/209 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0/212 (0) | 0/209 (0) | 1/212 (1) | 0/216 (0) | 0/209 (0)
Gout (Metabolism and nutrition disorders) | 0/212 (0) | 0/209 (0) | 3/212 (3) | 1/216 (1) | 0/209 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0/212 (0) | 1/209 (1) | 1/212 (1) | 0/216 (0) | 1/209 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 1/209 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 2/209 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1/212 (1) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Obesity (Metabolism and nutrition disorders) | 1/212 (1) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Podagra (Metabolism and nutrition disorders) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 1/209 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0/212 (0) | 0/209 (0) | 1/212 (1) | 0/216 (0) | 1/209 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0/212 (0) | 1/209 (1) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1/212 (1) | 3/209 (3) | 2/212 (3) | 10/216 (10) | 11/209 (13)
Bone pain (Musculoskeletal and connective tissue disorders) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 1/209 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 1/209 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 1/216 (1) | 0/209 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 2/216 (2) | 0/209 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0/212 (0) | 1/209 (1) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 1/209 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 1/209 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0/212 (0) | 2/209 (2) | 0/212 (0) | 2/216 (2) | 5/209 (6)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1/212 (1) | 0/209 (0) | 0/212 (0) | 1/216 (1) | 0/209 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2/212 (2) | 0/209 (0) | 1/212 (1) | 0/216 (0) | 1/209 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0/212 (0) | 1/209 (1) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0/212 (0) | 3/209 (4) | 3/212 (3) | 6/216 (6) | 6/209 (7)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0/212 (0) | 0/209 (0) | 1/212 (1) | 0/216 (0) | 0/209 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0/212 (0) | 3/209 (5) | 5/212 (5) | 2/216 (2) | 3/209 (3)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0/212 (0) | 0/209 (0) | 1/212 (1) | 0/216 (0) | 0/209 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1/212 (1) | 1/209 (1) | 1/212 (1) | 0/216 (0) | 0/209 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1/212 (1) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 1/209 (1)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 1/209 (1)
Burning sensation (Nervous system disorders) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 1/216 (1) | 1/209 (1)
Dizziness (Nervous system disorders) | 1/212 (1) | 0/209 (0) | 1/212 (1) | 1/216 (1) | 3/209 (3)
Headache (Nervous system disorders) | 6/212 (6) | 5/209 (5) | 6/212 (7) | 11/216 (11) | 7/209 (8)
Hypoaesthesia (Nervous system disorders) | 0/212 (0) | 0/209 (0) | 1/212 (1) | 0/216 (0) | 0/209 (0)
Lethargy (Nervous system disorders) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 1/216 (1) | 0/209 (0)
Nerve compression (Nervous system disorders) | 1/212 (1) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Neuralgia (Nervous system disorders) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 1/209 (1)
Neuropathy peripheral (Nervous system disorders) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 1/209 (1)
Paraesthesia (Nervous system disorders) | 0/212 (0) | 1/209 (1) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Sciatica (Nervous system disorders) | 0/212 (0) | 0/209 (0) | 1/212 (1) | 0/216 (0) | 1/209 (1)
Somnolence (Nervous system disorders) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 1/209 (1)
Syncope (Nervous system disorders) | 0/212 (0) | 2/209 (3) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Anxiety (Psychiatric disorders) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 1/216 (1) | 0/209 (0)
Depression (Psychiatric disorders) | 0/212 (0) | 1/209 (1) | 2/212 (2) | 1/216 (1) | 0/209 (0)
Insomnia (Psychiatric disorders) | 1/212 (1) | 0/209 (0) | 0/212 (0) | 2/216 (2) | 0/209 (0)
Sleep disorder (Psychiatric disorders) | 0/212 (0) | 1/209 (1) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Bladder spasm (Renal and urinary disorders) | 0/212 (0) | 1/209 (1) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Dysuria (Renal and urinary disorders) | 0/212 (0) | 1/209 (1) | 1/212 (1) | 0/216 (0) | 1/209 (1)
Nocturia (Renal and urinary disorders) | 0/212 (0) | 0/209 (0) | 1/212 (1) | 1/216 (1) | 1/209 (1)
Pollakiuria (Renal and urinary disorders) | 0/212 (0) | 0/209 (0) | 1/212 (1) | 0/216 (0) | 1/209 (1)
Renal cyst (Renal and urinary disorders) | 0/212 (0) | 1/209 (1) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Urinary hesitation (Renal and urinary disorders) | 0/212 (0) | 1/209 (1) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Urine flow decreased (Renal and urinary disorders) | 0/212 (0) | 0/209 (0) | 1/212 (1) | 0/216 (0) | 0/209 (0)
Balanitis (Reproductive system and breast disorders) | 0/212 (0) | 0/209 (0) | 1/212 (1) | 0/216 (0) | 0/209 (0)
Breast pain (Reproductive system and breast disorders) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 1/216 (2) | 0/209 (0)
Gynaecomastia (Reproductive system and breast disorders) | 1/212 (1) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Painful erection (Reproductive system and breast disorders) | 0/212 (0) | 1/209 (1) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 1/216 (1) | 0/209 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1/212 (1) | 3/209 (3) | 2/212 (2) | 2/216 (2) | 0/209 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0/212 (0) | 1/209 (1) | 2/212 (2) | 0/216 (0) | 1/209 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0/212 (0) | 2/209 (2) | 2/212 (2) | 1/216 (1) | 0/209 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0/212 (0) | 0/209 (0) | 2/212 (2) | 2/216 (2) | 0/209 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0/212 (0) | 1/209 (1) | 0/212 (0) | 0/216 (0) | 1/209 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1/212 (1) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 1/209 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0/212 (0) | 1/209 (1) | 1/212 (1) | 0/216 (0) | 0/209 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0/212 (0) | 1/209 (1) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2/212 (2) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0/212 (0) | 1/209 (1) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0/212 (0) | 0/209 (0) | 1/212 (1) | 0/216 (0) | 0/209 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0/212 (0) | 1/209 (1) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0/212 (0) | 0/209 (0) | 1/212 (4) | 0/216 (0) | 1/209 (1)
Rash (Skin and subcutaneous tissue disorders) | 1/212 (1) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 2/209 (2)
Skin irritation (Skin and subcutaneous tissue disorders) | 2/212 (2) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Carpal tunnel decompression (Surgical and medical procedures) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 0/216 (0) | 1/209 (1)
Dental operation (Surgical and medical procedures) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 1/216 (1) | 0/209 (0)
Sinus operation (Surgical and medical procedures) | 0/212 (0) | 1/209 (1) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Tooth extraction (Surgical and medical procedures) | 0/212 (0) | 1/209 (1) | 1/212 (1) | 0/216 (0) | 1/209 (1)
Umbilical hernia repair (Surgical and medical procedures) | 0/212 (0) | 0/209 (0) | 0/212 (0) | 1/216 (1) | 0/209 (0)
Blood pressure fluctuation (Vascular disorders) | 0/212 (0) | 0/209 (0) | 1/212 (1) | 0/216 (0) | 0/209 (0)
Flushing (Vascular disorders) | 0/212 (0) | 1/209 (1) | 0/212 (0) | 0/216 (0) | 0/209 (0)
Hot flush (Vascular disorders) | 0/212 (0) | 0/209 (0) | 1/212 (1) | 0/216 (0) | 0/209 (0)
Hypertension (Vascular disorders) | 1/212 (1) | 0/209 (0) | 4/212 (4) | 1/216 (1) | 0/209 (0)
Hypotension (Vascular disorders) | 0/212 (0) | 0/209 (0) | 1/212 (1) | 0/216 (0) | 0/209 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days